CLINICAL TRIAL: NCT02748811
Title: Effect of Geriatric Intervention in Frail Elderly Patients Receiving Chemotherapy for Colorectal Cancer
Acronym: GERICO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Danish Cancer Society (Other)
Responsible Party: Principal Investigator, Cecilia Lund, MD, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: GERICO
Record Dates: First submitted 2016-03-31; First posted 2016-04-22 (Estimated); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Colorectal Neoplasms
Keywords: elderly; intervention study; geriatrics; chemotherapy
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (No Intervention): The control group receives standard treatment with 6 months of adjuvant chemotherapy or first -line chemotherapy until operation, other scheduled change in treatment or progression. If the patient has other health problems, those issues will be assessed either by the oncologist or by the general practitioner. Validated quality of life questionnaires will be filled in prior to start, after 2 months and at the end of treatment.
- Intervention group (Active Comparator): The intervention group also receives standard treatment with 6 months of adjuvant chemotherapy or first -line chemotherapy until operation, other scheduled change of treatment or progression. They will simultaneously receive full geriatric assessement and intervention. The clinical examination includes laboratory parameters, review of medication list, psycho-cognitive assessement, screening for malnutrition and need of physiotherapy, optimizing social support. Validated quality of life questionnaires will be filled in prior to start, after 2 months and at the end of treatment.
  Interventions: Other: Intervention group

INTERVENTIONS:
Other: Intervention group — The intervention group also receives standard treatment with 6 months of adjuvant chemotherapy or first -line chemotherapy until operation, other scheduled change of treatment or progression. The participants will simultaneously receive full geriatric assessement and intervention. The clinical examination includes laboratory parameters, review of medication list, psycho-cognitive assessement, screening for malnutrition and need of physiotherapy, optimizing social support. Validated quality of life questionnaires will be filled in prior to start, after 2 months and at the end of treatment.
  Other Names: Comprehensive geriatric assessement and intervention
  Arms: Intervention group

SUMMARY:
GERICO is a randomized, controlled prospective trial. The aim is to investigate if frail, elderly patients with stage II-IV colorectal cancer, will profit from full comprehensive geriatric assessment and intervention before and during treatment with chemotherapy.

The hypotheses are: Optimizing the health conditions and functional status of frail elderly patients who suffers from stage II-IV colorectal cancer, with geriatric intervention will lead to a higher grade of completing the planned chemotherapy and at higher dose intensity. This will also result in a higher overall survival and improve quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Frail according to the screening tool G8 ( ≤14 / 17points)
* Performance status 0-2 and life expectancy ≥ 3 months
* Patients who have undergone surgery for stage III / high-risk stage II colorectal cancer or patients with unresectable or metastatic disease
* Are assessed to receive adjuvant chemotherapy or first -line chemotherapy
* Meets the criteria to receive preventive chemotherapy with 5-FU or capecitabine +/- oxaliplatin or first -line chemotherapy with 5-FU / irinotecan and / or oxaliplatin , capecitabine +/- possibly with the addition of immunotherapy in the form of cetuximab , panitumumab or bevacizumab.
* Informed written and oral consent

Exclusion Criteria:

* Other malignancy except basal cell carcinoma and squamous cell carcinoma in situ cervicis uteri in 5 years
* Patients in simultaneously drug trials
* The patient must not have previously received adjuvant chemotherapy in the GERICO Protocol

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 140 (Actual)
Dates: Start 2015-05; Primary Completion 2019-09 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
Number of patients completing planned treatment without dose reductions | 12 month after randomization

SECONDARY OUTCOMES:
Occurrence of dose reductions | 1 month after end of treatment
  Data will be collected by reviewing patients medical charts
delay of treatment | 1 month after end of treatment
  Data will be collected by reviewing patients medical charts
Adverse events to treatment | 1 month after end of treatment
  Adverse events will be registered for every cycle of treatment and assessed by an oncologist according to CTC- criteria version 4.0.
time to recurrence | up to 80 months
  Data will be collected by reviewing patients medical charts
Survival | up to 80 months
  Data will be collected by reviewing patients medical charts
Cancer specific mortality | up to 80 months
  Data will be collected by reviewing patients medical charts
Quality of Life prior | at 0 months and after 2 months and at the end of the treatment;e.g. up to 12months.
  Quality of life questionnaires will be filled out by the participants

CONTACTS AND LOCATIONS:
Overall Officials: Cecilia M Lund, MD, Principal Investigator — Department of Oncology
Locations (1):
- Department of Oncology. Herlev and Gentofte Hospital, Herlev, Danmark, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lund CM, Vistisen KK, Olsen AP, Bardal P, Schultz M, Dolin TG, Ronholt F, Johansen JS, Nielsen DL. The effect of geriatric intervention in frail older patients receiving chemotherapy for colorectal cancer: a randomised trial (GERICO). Br J Cancer. 2021 Jun;124(12):1949-1958. doi: 10.1038/s41416-021-01367-0. Epub 2021 Apr 7. PMID 33828260
- [Derived] Lund CM, Vistisen KK, Dehlendorff C, Ronholt F, Johansen JS, Nielsen DL. The effect of geriatric intervention in frail elderly patients receiving chemotherapy for colorectal cancer: a randomized trial (GERICO). BMC Cancer. 2017 Jun 28;17(1):448. doi: 10.1186/s12885-017-3445-8. PMID 28659138